CLINICAL TRIAL: NCT03338478
Title: Effect of Antiepileptic Drugs on Balance and Reaction Time
Brief Title: Balance and Anti-Epileptic Drugs
Acronym: AEDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erik J. Kobylarz (Other)
Collaborators: American Epilepsy Society (Other)
Responsible Party: Sponsor-Investigator, Erik J. Kobylarz, Fellow, GME Epilepsy, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D17186
Record Dates: First submitted 2017-10-20; First posted 2017-11-09 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epilepsy Patients (Experimental): Patients being tapered off of levetiracetam or lamotrigine monotherapy during epilepsy video monitoring. Patients will receive the Wii Balance Board and computerized reaction time testing.
  Interventions: Diagnostic Test: Wii Balance Board
- Healthy Control Group (Experimental): Patients without a diagnosis of epilepsy. Control participants will receive the Wii Balance Board and computerized reaction time testing.
  Interventions: Diagnostic Test: Wii Balance Board

INTERVENTIONS:
Diagnostic Test: Wii Balance Board — Participants will stand on the Wii Balance Board with eyes open, eyes closed, one two feet, and then standing on one leg at each study visit.

SUMMARY:
Patients with epilepsy exercise less than the general population. A barrier to exercise may be the effect of antiepileptic drugs on balance and reaction time. This proposal endeavors to study the effect of two common antiepileptic drugs (levetiracetam and lamotrigine) on balance and reaction time using a Wii balance board and reaction time test. This will be tested at descending doses in an epilepsy monitoring unit. Drug levels will be monitored, as well as center of pressure, and reaction time.

DETAILED DESCRIPTION:
Patients with epilepsy (PWE) exercise less compared to the general population. One barrier to participation in exercise is the subtle effect of anti epileptic drugs (AEDs) on balance and reaction time. Information on these measures in PWE is scarce, although previous data does suggest a detrimental effect. The objective of this trial is to study balance and reaction time in patients taking common AEDs. The investigators plan to study the effect of levetiracetam and lamotrigine on balance and reaction time. By studying patients in the epilepsy monitoring unit who are undergoing medication taper and withdrawal, the investigators can observe the effects of varying doses of these drugs within a single subject and also compare these data points to age matched controls. A Wii balance board (WBB) will be used to measure balance. It is hypothesized that levetiracetam and lamotrigine will elicit a dose-dependent, detrimental effect on balance and reaction time.

Patients admitted to the epilepsy monitoring unit who are currently taking levetiracetam or lamotrigine either in monotherapy will be recruited for the study. The target enrollment is 20 PWE, and 20 healthy controls.

For the PWE in the study, baseline AED blood levels will be obtained at baseline. The WBB has cells which detect load shifts in the body. Participants will stand on the WBB and remain as steady as possible. First on both feet with eyes open for 30 seconds, and then on both feet with eyes closed for 30 seconds, then on one foot with eyes open for 10 seconds, and then on one foot with eyes closed for 10 seconds. Each task will have 3 trials, with adequate break between.

Visit 2 will occur following weaning of AEDs. The investigators will measure center of pressure and reaction time testing similar to visit one. Blood AED levels will be checked at three half lives of the medication. This will be taken within 8 hours of visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Focal or generalized epilepsy
* On a stable dose of AEDs defined by no medication changes within the last month.
* On levetiracetam or lamotrigine monotherapy

Exclusion Criteria:

* Inability to stand independently for 30 seconds
* Peripheral neuropathy
* History of stroke or previous brain surgery
* Seizure within last 24 hours

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Balance | Up to six weeks.
  Balance measured by Wii Balance Board (WBB). The WBB has cells which detect load shifts in the body. Participants stand on both feet with eyes open; on both feet with eyes closed; on one foot with eyes open; and on one foot with eyes closed. Balancia software will be used to analyze the information.
Reaction Time | Up to six weeks.
  Participants will use dominant hand on mouse to click as quickly as possible in response to a prompt on a computer screen. Five trials will be conducted at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Kobylarz, M.D., PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data is not planned to be shared with outside researchers.